CLINICAL TRIAL: NCT07259421
Title: Survey of Practices Regarding the Use of Taurolidine Lock Solutions in Patients With Insertion of a Peripherally Inserted Central Catheter (PICC) in a Vascular Access Unit
Acronym: TAURO-USE2
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0315.
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Taurolidine Lock Solution
Keywords: vascular access unit; parenteral nutrition; peripherally inserted central catheter; catheter related infection; health care-associated infection; taurolidine; lock solution; survey of practices
MeSH Terms: conditions — Hyperphagia; Catheter-Related Infections; Cross Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to describe current practices regarding the administration of taurolidine lock solutions in relation to medical prescriptions for patients who have undergone peripherally inserted central catheter (PICC) implantation in the Vascular Access Unit as part of parenteral nutrition therapy. Our underlying hypothesis is that the use of taurolidine lock solutions may deviate from current recommendations, particularly with respect to administration procedures.

This study will allow us to characterize the use of taurolidine lock solutions in relation to medical prescriptions, identify potential deviations from recommended practices, and document any associated adverse events. It will also enable follow-up of PICC outcomes at 8 and 30 days after implantation in the Vascular Access Unit, whereas current follow-up is performed only at 8 days post-insertion.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has undergone PICC placement in the vascular access unit with an indication for parenteral nutrition supplementation.
* Patient not opposed to participating in this research.

Exclusion Criteria:

* Patient not speaking French
* Patient under guardianship or conservatorship
* Patient with major neurocognitive disorders
* Patient with severe hearing impairment
* Patient who do not have a telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion criteria will be recruited consecutively over a three-month period to minimize the risk of selection bias.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To characterize, through an assessment of current practices, the administration of taurolidine lock solutions as prescribed for patients who have undergone PICC implantation in the Vascular Access Unit as part of parenteral nutrition therapy. | Eight and thirty days after PICC placement in the Vascular Access Unit
  Proportion of patients with a prescription for a taurolidine lock solution who actually receive administrations of the prescribed lock solution (concordance between prescribed and administered product).
  Proportion of patients for whom lock solutions are administered in accordance with the manufacturer's instructions for use; compliant administration is defined as the nurse performing all recommended steps for applying the lock solution at the end of each parenteral nutrition infusion.
  Proportion of patients for whom lock solutions are withdrawn in accordance with the manufacturer's instructions for use (lock solutions aspirated before catheter use).
  Proportion of patients for whom lock solutions are disposed of in accordance with regulations for biological-hazard waste.

SECONDARY OUTCOMES:
Describe nurses' perceptions of their own knowledge regarding the use of taurolidine lock solutions. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Quantify, using a self-assigned score, nurses' level of knowledge concerning taurolidine lock solutions.
  Proportion of nurses aware of the various properties of lock solutions according to the references available on the market.
Describe the medical care provided by home service providers for patients receiving a PICC placement for parenteral nutrition supplementation. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and number of service providers working with patients at home.
Describe the supply chain for taurolidine lock solutions. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportions of procurement methods for taurolidine lock solutions for patients at home.
Describe the elements related to PICC placement. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportions of elements related to PICC placement: number of lumens, vein of insertion, side of insertion, duration of placement, and role of the inserter (nurse anesthetists or physician).
Characterize the functional status of the PICC over time. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Proportion of PICC in place and functional at 8 and 30 days post-insertion, defined as not requiring premature removal and allowing infusion and blood sampling.
Describe complications related to PICC placement. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportions of complications related to the PICC occurring within 8 and 30 days post-insertion.
Describe the causes of premature PICC removal. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportions of causes for premature PICC-line removal within 8 and 30 days post-insertion.
Describe adverse events related to the use of taurolidine lock solutions. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportion of adverse events potentially related to the use of a taurolidine lock solution, as reported by patients or healthcare providers.
Describe the difficulties encountered by healthcare professionals when using taurolidine lock solutions. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportion of difficulties encountered by home-care nurses when using taurolidine lock solutions.
Describe the information sources used by healthcare professionals regarding taurolidine lock solutions. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Nature and proportion of information sources consulted by nurses in the event of problems related to the use of a taurolidine lock solution or to the use of the PICC.
Characterize the use of device vigilance in the event of adverse events related to taurolidine lock solutions. | Eight and thirty days after PICC placement in the Vascular Access Unit.
  Proportion of nurses who would report to device vigilance any adverse events related to the use of a taurolidine lock solution or to the use of the PICC, should such events occur.

IPD SHARING:
Plan to Share IPD: No